CLINICAL TRIAL: NCT05164536
Title: Plasma P-tau2017 and Quantitative Amyloid PET Imaging in a Cognitively Normal Population
Brief Title: Plasma P-tau2017 and Quantitative Amyloid PET Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Plasma P-tau 2017
Record Dates: First submitted 2021-10-20; First posted 2021-12-20 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease
Keywords: AD
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]Florbetapir (Experimental): Participants will undergo amyloid PET imaging with an approved amyloid radiotracer (ie, [18F]Florbetapir (Amyvid™)) to assess β-amyloid neuritic plaque density.
  Interventions: Drug: Amyvid

INTERVENTIONS:
Drug: Amyvid — All participants will undergo a single β-amyloid PET scan with Amyvid.
  Other Names: [18F]Florbetapir

SUMMARY:
The overall goal of this protocol is to compare amyloid burden assessed by amyloid PET to plasma P-tau217 levels.

DETAILED DESCRIPTION:
The overall goal of this protocol is to compare amyloid burden assessed by amyloid PET to plasma P-tau217 levels. Other relevant AD-related investigational biomarkers may also be assessed in the provided samples. Apolipoprotein E (ApoE) genetic status will be evaluated with a serum sample.

ELIGIBILITY:
Inclusion Criteria (for all participants):

* Signed and dated written informed consent obtained from the subject.
* Male participants with partners of childbearing potential must commit to the use of 2 methods of contraception, one of which is a barrier method for male participants for the study duration.
* Male participants must not donate sperm for the study duration.
* Willing and able to cooperate with study procedures.
* Males and females.
* Participants aged ≥ 70, inclusive, at the time of Screening.
* Judged to be cognitively normal by an Investigator based on clinical judgment.

Exclusion Criteria (for all participants):

* Subject has received an investigational drug or device within 30 days of enrollment, unless in the opinion of the Investigator such medication or device will not impair subject safety or scientific integrity of the data.
* Contraindication to amyloid PET imaging or blood sampling.
* Have ever received an experimental or approved medication targeting amyloid or tau.
* Prior participation in other research protocols or clinical care in the last year that would result in radiation exposure exceeding the acceptable annual limit established by the U.S. Federal Guidelines (effective dose of 50 mSv, including the procedures in this clinical protocol).
* Pregnancy, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease that in the Investigator's judgment may interfere with the objectives of the study.
* Unsuitable veins for venipuncture.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Creation of a database of brain amyloid deposition by region using PET signal-to-noise ratio, SUVr . | 1 year
  Amyloid PET imaging will be used to measure regional brain amyloid deposition in each subject.

SECONDARY OUTCOMES:
Creation of a database of blood P-tau217 and other blood biomarkers. | 1 year
  Blood will be analyzed at Eli Lilly for P-tau217 and ApoE genotype. The analysis will be described in a separate analysis plan.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Information — http://invicro.com